CLINICAL TRIAL: NCT07327463
Title: Comparison of the Analgesic Efficacy of Ultrasound-guided Transversus Abdominis Plane Block and Single-dose Epidural Block in Patients Undergoing Umbilical Hernia Surgery.
Brief Title: Ultrasound-Guided Transversus Abdominis Plane Block Versus Epidural Block for Umbilical Hernia Analgesia
Status: Recruiting | Type: Observational
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Burçin Alaçam, MD, Anesthesiology Specialist, Sakarya University
Other Study IDs: SAU-ANE-BA-02
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Umbilical Hernia; Postoperative Pain Management
Keywords: Single-Dose Epidural Analgesia; Transversus Abdominis Plane Block; Postoperative Pain Management; Umbilical Hernia Surgery
MeSH Terms: conditions — Hernia, Umbilical | interventions — Anesthesia, Epidural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group Transversus Abdominis Plane Block: Patients in this group will undergo umbilical hernia surgery under general anesthesia. Following completion of the surgical procedure, postoperative analgesia will be provided using an ultrasound-guided transversus abdominis plane (TAP) block, performed according to routine clinical practice. The TAP block will be administered by an experienced anesthesiologist using standard techniques and local anesthetic agents. No additional interventions or investigational medications will be applied as part of the study.
  Postoperative pain intensity will be assessed using the Visual Analog Scale (VAS) at admission to and discharge from the post-anesthesia care unit, as well as at the 1st, 6th, 12th, and 24th postoperative hours. Rescue analgesia will be administered based on routine institutional protocols according to patient-reported pain scores.
  Interventions: Other: Ultrasound-Guided Transversus Abdominis Plane Block
- Group Single Dose Epidural Anesthesia: Patients in this group will undergo umbilical hernia surgery under single-dose epidural anesthesia administered as part of routine clinical practice. The epidural technique will be performed by an experienced anesthesiologist using standard institutional protocols. The single-dose epidural injection will be used to provide both intraoperative anesthesia and postoperative analgesia. No additional interventions or investigational medications will be administered for the purpose of this study.
  Postoperative pain intensity will be evaluated using the Visual Analog Scale (VAS) at admission to and discharge from the post-anesthesia care unit, as well as at the 1st, 6th, 12th, and 24th postoperative hours. Rescue analgesic treatment will be provided according to routine postoperative pain management protocols based on patient-reported pain scores.
  Interventions: Other: Single-Dose Epidural Anesthesia

INTERVENTIONS:
Other: Ultrasound-Guided Transversus Abdominis Plane Block — Ultrasound-guided transversus abdominis plane (TAP) block is performed as part of routine postoperative analgesia following general anesthesia in patients undergoing umbilical hernia surgery. The procedure is administered by an experienced anesthesiologist using standard institutional practice. No additional procedures or medications are applied specifically for the purpose of this observational study.
  Groups: Group Transversus Abdominis Plane Block
Other: Single-Dose Epidural Anesthesia — Single-dose epidural anesthesia is administered as part of routine clinical practice to provide intraoperative anesthesia and postoperative analgesia in patients undergoing umbilical hernia surgery. The technique is performed by an experienced anesthesiologist according to standard institutional protocols. No investigational interventions or study-specific modifications are implemented.
  Groups: Group Single Dose Epidural Anesthesia

SUMMARY:
This observational study aims to compare the postoperative analgesic effectiveness of ultrasound-guided transversus abdominis plane (TAP) block and single-dose epidural anesthesia in patients undergoing umbilical hernia surgery. Pain intensity will be assessed using the Visual Analog Scale (VAS) at predefined postoperative time points. The study seeks to determine which analgesic approach provides superior pain control and patient satisfaction in the postoperative period.

DETAILED DESCRIPTION:
Postoperative pain management plays a critical role in reducing the adverse consequences of surgery, facilitating early mobilization, enhancing patient comfort, and promoting rapid recovery and discharge. Epidural analgesia is widely regarded as the gold standard for postoperative pain control due to its strong analgesic efficacy and its ability to reduce the need for additional anesthetic and analgesic agents. However, peripheral and fascial plane blocks such as the transversus abdominis plane (TAP) block have gained increasing popularity because of their opioid-sparing effects and favorable side-effect profiles.

The transversus abdominis plane is a neurofascial plane located between the internal oblique and transversus abdominis muscles and provides somatic analgesia to the anterolateral abdominal wall by blocking the thoracolumbar nerves from T9 to L1. Previous studies have demonstrated that TAP block is associated with reduced postoperative pain scores, decreased opioid consumption, and fewer opioid-related adverse effects.

This study is designed as an observational comparison of two routinely applied analgesic strategies in patients undergoing umbilical hernia surgery. Patients aged between 18 and 65 years, classified as American Society of Anesthesiologists (ASA) physical status I or II, will be included. Depending on the anesthesiologist's clinical judgment and routine practice, patients undergo surgery either under single-dose epidural anesthesia or under general anesthesia followed by postoperative ultrasound-guided TAP block for analgesia.

No additional interventions or medications will be administered for the purpose of this study. Data collection will begin once patients are admitted to the postoperative recovery unit. Postoperative pain intensity will be assessed using the Visual Analog Scale (VAS) at recovery room admission and discharge, as well as at the 1st, 6th, 12th, and 24th postoperative hours. Rescue analgesia will be administered according to routine clinical protocols based on patients' reported pain levels.

The primary objective of this study is to compare the analgesic effectiveness of single-dose epidural anesthesia and TAP block in umbilical hernia surgery. Secondary objectives include the evaluation of patient satisfaction and the identification of the most effective postoperative analgesic approach within routine clinical practice. As all procedures involved are part of standard care, this study does not constitute an interventional drug trial but rather an observational assessment of established analgesic techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 65 years
* Patients scheduled for elective umbilical hernia surgery
* ASA physical status I or II
* Patients who undergo surgery under either: Single-dose epidural anesthesia, or general anesthesia with postoperative ultrasound-guided transversus abdominis plane (TAP) block, as part of routine clinical practice
* Ability to understand and use the Visual Analog Scale (VAS)
* Provision of written informed consent

Exclusion Criteria:

* ASA physical status III or higher
* Known allergy or contraindication to local anesthetic agents
* Coagulopathy or ongoing anticoagulant/antiplatelet therapy contraindicating regional anesthesia
* Infection at the site of epidural or TAP block application
* History of chronic pain, long-term opioid use, or chronic analgesic consumption
* Neurological disorders affecting pain perception or assessment
* Severe hepatic or renal disease
* Pregnancy or lactation
* Inability to cooperate with postoperative pain assessment or inability to use VAS
* Emergency surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 to 65 years with American Society of Anesthesiologists (ASA) physical status I or II who are scheduled to undergo elective umbilical hernia surgery. Patients included in the study receive anesthesia and postoperative analgesia as part of routine clinical practice, either with single-dose epidural anesthesia or with general anesthesia followed by ultrasound-guided transversus abdominis plane (TAP) block.
  All patients are managed according to standard institutional surgical and anesthetic protocols. No additional interventions, medications, or procedures are performed for research purposes. Postoperative pain assessment is conducted using the Visual Analog Scale (VAS) during the postoperative period. The study population reflects real-world clinical practice in umbilical hernia surgery.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-01-15 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Visuel Analog Scale 6th hour | postoperative 6th hour
  Postoperative pain intensity will be evaluated using the Visual Analog Scale (VAS) at the 6th postoperative hour to compare the analgesic effectiveness of single-dose epidural anesthesia and ultrasound-guided transversus abdominis plane (TAP) block. The Visual Analog Scale (VAS) is used to assess pain intensity on a numeric scale ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst pain imaginable. Patients are asked to select the number that best represents their current level of pain at the time of assessment. Increasing scores reflect increasing pain severity, with values of 1-3 considered mild pain, 4-6 moderate pain, and 7-10 severe pain. The VAS is a simple, reliable, and sensitive tool for detecting changes in pain intensity over time and is widely used in clinical trials and postoperative pain assessment.

SECONDARY OUTCOMES:
Visuel Analog Scale 30.minutes | postoperative 30.minutes
  Postoperative pain intensity will be evaluated using the Visual Analog Scale (VAS) at the 30 minute after postoperative hour to compare the analgesic effectiveness of single-dose epidural anesthesia and ultrasound-guided transversus abdominis plane (TAP) block. The Visual Analog Scale (VAS) is used to assess pain intensity on a numeric scale ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst pain imaginable. Patients are asked to select the number that best represents their current level of pain at the time of assessment. Increasing scores reflect increasing pain severity, with values of 1-3 considered mild pain, 4-6 moderate pain, and 7-10 severe pain. The VAS is a simple, reliable, and sensitive tool for detecting changes in pain intensity over time and is widely used in clinical trials and postoperative pain assessment.
Visuel Analog Scale 1st hour | postoperartive 1st hour
  Postoperative pain intensity will be evaluated using the Visual Analog Scale (VAS) at the 1st postoperative hour to compare the analgesic effectiveness of single-dose epidural anesthesia and ultrasound-guided transversus abdominis plane (TAP) block. The Visual Analog Scale (VAS) is used to assess pain intensity on a numeric scale ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst pain imaginable. Patients are asked to select the number that best represents their current level of pain at the time of assessment. Increasing scores reflect increasing pain severity, with values of 1-3 considered mild pain, 4-6 moderate pain, and 7-10 severe pain. The VAS is a simple, reliable, and sensitive tool for detecting changes in pain intensity over time and is widely used in clinical trials and postoperative pain assessment.
Visuel Analog Scale 2nd hour | postoperative 2nd hour
  Postoperative pain intensity will be evaluated using the Visual Analog Scale (VAS) at the 2nd postoperative hour to compare the analgesic effectiveness of single-dose epidural anesthesia and ultrasound-guided transversus abdominis plane (TAP) block. The Visual Analog Scale (VAS) is used to assess pain intensity on a numeric scale ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst pain imaginable. Patients are asked to select the number that best represents their current level of pain at the time of assessment. Increasing scores reflect increasing pain severity, with values of 1-3 considered mild pain, 4-6 moderate pain, and 7-10 severe pain. The VAS is a simple, reliable, and sensitive tool for detecting changes in pain intensity over time and is widely used in clinical trials and postoperative pain assessment.
Visuel Analog Scale 12th hour | postoperative 12th hour
  Postoperative pain intensity will be evaluated using the Visual Analog Scale (VAS) at the 12th postoperative hour to compare the analgesic effectiveness of single-dose epidural anesthesia and ultrasound-guided transversus abdominis plane (TAP) block. The Visual Analog Scale (VAS) is used to assess pain intensity on a numeric scale ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst pain imaginable. Patients are asked to select the number that best represents their current level of pain at the time of assessment. Increasing scores reflect increasing pain severity, with values of 1-3 considered mild pain, 4-6 moderate pain, and 7-10 severe pain. The VAS is a simple, reliable, and sensitive tool for detecting changes in pain intensity over time and is widely used in clinical trials and postoperative pain assessment.
Visuel Analog Scale 24th hour | postoperative 24th hour
  Postoperative pain intensity will be evaluated using the Visual Analog Scale (VAS) at the 24th postoperative hour to compare the analgesic effectiveness of single-dose epidural anesthesia and ultrasound-guided transversus abdominis plane (TAP) block. The Visual Analog Scale (VAS) is used to assess pain intensity on a numeric scale ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst pain imaginable. Patients are asked to select the number that best represents their current level of pain at the time of assessment. Increasing scores reflect increasing pain severity, with values of 1-3 considered mild pain, 4-6 moderate pain, and 7-10 severe pain. The VAS is a simple, reliable, and sensitive tool for detecting changes in pain intensity over time and is widely used in clinical trials and postoperative pain assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University-Anesthesiology and Reanimation Department, Sakarya, Serdivan, Turkey (Türkiye)

REFERENCES:
- [Result] Yadav U, Doneria D, Gupta V, Verma S. Ultrasound-Guided Transversus Abdominis Plane Block Versus Single-Shot Epidural Block for Postoperative Analgesia in Patients Undergoing Inguinal Hernia Surgery. Cureus. 2023 Jan 17;15(1):e33876. doi: 10.7759/cureus.33876. eCollection 2023 Jan. PMID 36819433